CLINICAL TRIAL: NCT00156741
Title: IntAct, Study on Promotion of Intrinsic Activity.
Brief Title: Efficacy of a Pacemaker Algorithm in Promotion of the Intrinsic Heart Activity.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medtronic BRC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CMD 287
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2005-09

CONDITIONS: Bradycardia; Sick Sinus Syndrome, AV Block
Keywords: Refined ventricular pacing
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Atrioventricular Block

INTERVENTIONS:
Device: Vitatron C50 D Model C50A2 of Vitatron C60 DR model C60A2
Procedure: Required pacemaker setting

SUMMARY:
The purpose of this study is to provide evidence that the Refined Ventricular Pacing Algorithm leads to clinically relevant reduction (at least 50% reduction) of the incidence of ventricular pacing.

DETAILED DESCRIPTION:
Electrical stimulation in the apex of the right ventricle ( ventricular pacing) usually improves the heart function of patients with a pacemaker and can even be life-saving. However, evidence is accumulating that ventricular pacing may also have undesired long-term cardiac effects. Therefore, it makes sense to limit ventricular pacing to the absolute required minimum. The functionality RVP (Refined Ventricular Pacing) in the C-series 2nd generation pacemakers of Vitatron B.V. Arnhem, the Netherlands is designed to reduce ventricular pacing.

After implantation of the Vitatron C50 D model C50A2 (pacemaker) or Vitatron C60 DR model C60A2 (pacemaker) and a 4-6 weeks stabilization period, proper functioning of pacemaker and leads (stimulation- and sensing parameters) is checked. The pacemakers will be programmed according to predefined settings.

In the following 4-weeks Baseline period diagnostic data (atrial fibrillation burden and percentage of ventricular pacing (% VP)) are collected in the pacemaker memory. Based on these data, patients will be excluded from further participation (patients with more than 15% atrial fibrillation) or subdivided into three groups: (a) < 30% VP (30- VP group), (b) >30% VP, Sick Sinus Syndrome and normal conductivity (SSS group), (c) >30% VP, 1st or 2nd degree AV block. Patients in these three groups will be treated for 4 weeks alternatively with the RVP functionality switched ON or OFF. The order will be determined by randomization. At the end of these two cross-over periods the % VP and the judgment of the patients of the last period will be assessed. Adverse events will be recorded from the moment of study enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Patients shall be willing to sign the Patient Informed Consent for this study
* Patients shall have at least one of the following indications for a pacemaker: - Sick Sinus Syndrome with normal QRS complexes
* First degree AV block with a PR interval <_220 ms for patients <_ 70 years of age, or <_ 260 for patients over 70 years
* Second-degree AV block, mobitz I (wenckebach) or mobitz II
* Patients shall be available for follow-up for the duration of their participation.

Exclusion Criteria:

* Patients involved in another investigation study conducted in parallel to this study
* Patients younger than 18 years of age and/or patients that do NOT meet other local requirements for participation
* Pregnant patients
* Patients with lead integrity problems (and the lead is not being replaced)
* Patients with persistant AF
* Patients with a complete AV block
* Patients with NYHA (New York Heart Association0 class III and IV
* Patients who underwent thoracic surgery in the last three months or are expected to have in the near future
* Patients with a 2:1 block
* Patients with a life expectancy less than half a year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Calculation of reduction in % VP when RVP algorithm is ON versus OFF, recording % VP at 4 and 8 weeks after randomization

SECONDARY OUTCOMES:
Occurrence of possible undesired consequences of the RVP algorithm (e.g. retrograde conduction; AF burden) and adverse events in the periods with the algorithm switched ON versus OFF, 4 and 8 weeks after randomization
Patient's opinion about treatment (on a six-point scale), at 4 and 8 weeks after randomization
explorative subanalysis on patients with different arrhythmias and/or conducting system defects to investigate in which type of patients the RVP algorithm will have the largest impact on %VP
Reproducibility of the %VP assessment, comparison %VP during Baseline periode and 4-week study period with RVP OFF

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Binner, MD, Study Chair — Universitätsklinikum Ulm, Ulm, Germany; Chris van Groeningen, MD, Study Director — Vitatron B.V., Arnhem, The Netherlands
Locations (30):
- A.ö. Krankenhaus der Elisabethinen Linz, Linz, Austria
- Czechia (6):
  - Fakultni nemocnice u svate Anny v Berne, Brno
  - Fakulti Nemocnice, University Hospital of Brno-Bohunice, Brno-Bohunice
  - University Hospital with Polyclinics Ostrava, Ostrava
  - Kardiologicka kllinika, Prague
  - Nemocnice Na Homolce Hospital, Prague
  - Masarykova Nemocnice, Ústí nad Labem
- Denmark (2):
  - Hillerod Sygehus, Hillerød
  - Vejle Sygehus, Vejle
- Finland (2):
  - Tampere University Central Hospital, Tampere
  - University of Oulu, Depart. of Internal Medicine, Div. of Cardiology, University of Oulu
- Germany (6):
  - Elisabeth Krankenhaus, Essen
  - Stadt. Klinikum Leverkussen, Leverkussen
  - Deutschen Herzzentrum Munchen des Freistaates Bayern Klinik an der TU Munchen, München
  - Stadtisches Klinikum Pforzheim, Pforazheim
  - Kreiskrankenhaus Rottweil, Rottweil
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Arcispedale S. Maria Nuova, Reggio Emilia, Emilia-Romagna
  - San Camillo De' Lellis, Rieti
- Netherlands (4):
  - Meander Medisch Centrum, Lokatie Lichtenberg, Amersfoort
  - St. Lucas Andreas Ziekenhuis, Amsterdam
  - Catharina Hospital, Eindhoven
  - Bronovo Ziekenhuis, The Hague
- Russia (2):
  - Hospital Nr.: 26, Saint Petersburg
  - Pokrovskiy Hospital, Saint Petersburg
- Sweden (2):
  - Medicinkliniken, Borås
  - Karolinska University Hospital Hjartkliniken, Stockholm
- Switzerland (2):
  - Kantonsspital Kardiologie, Basel
  - Inselspital Bern, Schweizer Herz- und Gefasszentrum, Bern
- Blackpool Victoria Hospital, Blackpool, United Kingdom

REFERENCES:
- [Background] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Background] Skanes AC, Krahn AD, Yee R, Klein GJ, Connolly SJ, Kerr CR, Gent M, Thorpe KE, Roberts RS; Canadian Trial of Physiologic Pacing. Progression to chronic atrial fibrillation after pacing: the Canadian Trial of Physiologic Pacing. CTOPP Investigators. J Am Coll Cardiol. 2001 Jul;38(1):167-72. doi: 10.1016/s0735-1097(01)01326-2. PMID 11451268
- [Background] Gillis AM, Goldman BS, Yee R, Irwin ME, Wilson SL, Ashton T, Philippon F, Fraser JD, Clavette P, Tyers GF. Cardiac pacing in Canada in 1998: working towards optimal pacing therapy. Canadian Working Group on Cardiac Pacing. Can J Cardiol. 1998 Sep;14(9):1115-20. PMID 9779016
- [Background] Lamas GA, Orav EJ, Stambler BS, Ellenbogen KA, Sgarbossa EB, Huang SK, Marinchak RA, Estes NA 3rd, Mitchell GF, Lieberman EH, Mangione CM, Goldman L. Quality of life and clinical outcomes in elderly patients treated with ventricular pacing as compared with dual-chamber pacing. Pacemaker Selection in the Elderly Investigators. N Engl J Med. 1998 Apr 16;338(16):1097-104. doi: 10.1056/NEJM199804163381602. PMID 9545357
- [Background] Danish pacemaker and ICD register. 1999. Pacing Clin Electrophysiol. 2000 Oct;23(10 Pt 2):S1-93. No abstract available. PMID 11758538
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Background] The MOST Trial Investigators. Effect of pacing mode and cumulative percent time ventricular paced on heart failure in patients with sick sinus syndrome and baseline QRS duration < 120 milliseconds in MOST. PACE 2002; 561 Abstract 155.
- [Background] The MOST Trial Investigators. Baseline QRS duration ≥ 120 milliseconds and cumulative percent time ventricular paced predicts increased risk of heart failure, stroke and death in DDDR-paced patients with sick sinus syndrome in MOST. PACE 2002; 690 Abstract 672
- [Background] International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals. N Engl J Med. 1991 Feb 7;324(6):424-8. doi: 10.1056/NEJM199102073240624. No abstract available. PMID 1987468
- [Background] Andersen HR, Thuesen L, Bagger JP, Vesterlund T, Thomsen PE. Prospective randomised trial of atrial versus ventricular pacing in sick-sinus syndrome. Lancet. 1994 Dec 3;344(8936):1523-8. doi: 10.1016/s0140-6736(94)90347-6. PMID 7983951
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Kristensen L, Nielsen JC, Mortensen PT, Pedersen OL, Pedersen AK, Andersen HR. Incidence of atrial fibrillation and thromboembolism in a randomised trial of atrial versus dual chamber pacing in 177 patients with sick sinus syndrome. Heart. 2004 Jun;90(6):661-6. doi: 10.1136/hrt.2003.016063. PMID 15145874
- [Background] Barold SS. Indications for permanent cardiac pacing in first-degree AV block: class I, II, or III? Pacing Clin Electrophysiol. 1996 May;19(5):747-51. doi: 10.1111/j.1540-8159.1996.tb03355.x. No abstract available. PMID 8734740
- [Background] Bode F, Wiegand U, Katus HA, Potratz J. Inhibition of ventricular stimulation in patients with dual chamber pacemakers and prolonged AV conduction. Pacing Clin Electrophysiol. 1999 Oct;22(10):1425-31. doi: 10.1111/j.1540-8159.1999.tb00345.x. PMID 10588143
- [Background] Boute W, Brunekreeft W. AV delay hysteresis in dual chamber pacing: initial results from the Ruby Clinical Investigation. Vitatext 1994; 1: 13-14
- [Background] Brandt J, Anderson H, Fahraeus T, Schuller H. Natural history of sinus node disease treated with atrial pacing in 213 patients: implications for selection of stimulation mode. J Am Coll Cardiol. 1992 Sep;20(3):633-9. doi: 10.1016/0735-1097(92)90018-i. PMID 1512343
- [Background] Carisma MB, Manalo JM, Chua WT. Atrioventricular conduction in sick sinus syndrome. Pacing Clin Electrophysiol. 1988 Nov;11(11 Pt 2):1636-40. doi: 10.1111/j.1540-8159.1988.tb06287.x. PMID 2463525
- [Background] Charles RG, McComb JM. Systematic trial of pacing to prevent atrial fibrillation (STOP-AF). Heart. 1997 Sep;78(3):224-5. doi: 10.1136/hrt.78.3.224. No abstract available. PMID 9391281
- [Background] Cohen SI, Frank HA. Preservation of active atrial transport; an important clinical consideration in cardiac pacing. Chest. 1982 Jan;81(1):51-4. doi: 10.1378/chest.81.1.51. PMID 7053943
- [Background] Connolly SJ, Talajic M, Roy D, Tang ASL, Lav C, Bonilla L, Gillis AM. The effect of pacemaker selection on functional capacity in the Canadian Trial of Physiologic Pacing (CTOPP). Circulation 1999; 100(suppl I): I-465
- [Background] Clarke KW, Connelly DT, Charles RG. Single chamber atrial pacing: an underused and cost-effective pacing modality in sinus node disease. Heart. 1998 Oct;80(4):387-9. doi: 10.1136/hrt.80.4.387. PMID 9875119
- [Background] Elshot SR, el Gamal MI, Tielen KH, van Gelder BM. Incidence of atrioventricular block and chronic atrial flutter/fibrillation after implantation of atrial pacemakers; follow-up of more than ten years. Int J Cardiol. 1993 Mar;38(3):303-8. doi: 10.1016/0167-5273(93)90249-g. PMID 8463012
- [Background] Grimm W, Langenfeld H, Maisch B, Kochsiek K. Symptoms, cardiovascular risk profile and spontaneous ECG in paced patients: a five-year follow-up study. Pacing Clin Electrophysiol. 1990 Dec;13(12 Pt 2):2086-90. doi: 10.1111/j.1540-8159.1990.tb06947.x. PMID 1704598
- [Background] Harper GR, Pina IL, Kutalek SP. Intrinsic conduction maximizes cardiopulmonary performance in patients with dual chamber pacemakers. Pacing Clin Electrophysiol. 1991 Nov;14(11 Pt 2):1787-91. doi: 10.1111/j.1540-8159.1991.tb02767.x. PMID 1721176
- [Background] Haywood GA, Ward J, Ward DE, Camm AJ. Atrioventricular Wenckebach point and progression to atrioventricular block in sinoatrial disease. Pacing Clin Electrophysiol. 1990 Dec;13(12 Pt 2):2054-8. doi: 10.1111/j.1540-8159.1990.tb06941.x. PMID 1704592
- [Background] Hesselson AB, Parsonnet V, Bernstein AD, Bonavita GJ. Deleterious effects of long-term single-chamber ventricular pacing in patients with sick sinus syndrome: the hidden benefits of dual-chamber pacing. J Am Coll Cardiol. 1992 Jun;19(7):1542-9. doi: 10.1016/0735-1097(92)90616-u. PMID 1593051
- [Background] Jutzy RV, Feenstra L, Pai R, Florio J, Bansal R, Aybar R, Levine PA. Comparison of intrinsic versus paced ventricular function. Pacing Clin Electrophysiol. 1992 Nov;15(11 Pt 2):1919-22. doi: 10.1111/j.1540-8159.1992.tb02994.x. PMID 1279572
- [Background] Kallryd A, Kruse I, Ryden L. Atrial inhibited pacing in the sick sinus node syndrome: clinical value and the demand for rate responsiveness. Pacing Clin Electrophysiol. 1989 Jun;12(6):954-61. doi: 10.1111/j.1540-8159.1989.tb05033.x. PMID 2472623
- [Background] Kerr CR, Tyers GF, Vorderbrugge S. Atrial pacing: efficacy and safety. Pacing Clin Electrophysiol. 1989 Jul;12(7 Pt 1):1049-54. doi: 10.1111/j.1540-8159.1989.tb01925.x. PMID 2476740
- [Background] Kristensen L, Nielsen JC, Andersen HR. Outcome of patients with sick sinus syndrome treated by different pacing modalities. In Ovsyshcher IE (ed): Cardiac arrhythmias and device therapy results and perspectives for the new century. Futura Publishing Company Inc., Armonk NY, 2000, 323-332.
- [Background] Leclercq C, Gras D, Le Helloco A, Nicol L, Mabo P, Daubert C. Hemodynamic importance of preserving the normal sequence of ventricular activation in permanent cardiac pacing. Am Heart J. 1995 Jun;129(6):1133-41. doi: 10.1016/0002-8703(95)90394-1. PMID 7754944
- [Background] Mattioli AV, Vivoli D, Mattioli G. Influence of pacing modalities on the incidence of atrial fibrillation in patients without prior atrial fibrillation. A prospective study. Eur Heart J. 1998 Feb;19(2):282-6. doi: 10.1053/euhj.1997.0616. PMID 9519322
- [Background] Montanez A, Hennekens CH, Zebede J, Lamas GA. Pacemaker mode selection: the evidence from randomized trials. Pacing Clin Electrophysiol. 2003 May;26(5):1270-82. doi: 10.1046/j.1460-9592.2003.t01-1-00179.x. PMID 12765457
- [Background] Narula OS. Atrioventricular conduction defects in patients with sinus bradycardia. Analysis by His bundle recordings. Circulation. 1971 Dec;44(6):1096-110. doi: 10.1161/01.cir.44.6.1096. No abstract available. PMID 5127836
- [Background] Nielsen JC, Pedersen AK, Mortensen PT, Andersen HR. Programming a fixed long atrioventricular delay is not effective in preventing ventricular pacing in patients with sick sinus syndrome. Europace. 1999 Apr;1(2):113-20. doi: 10.1053/eupc.1998.0026. PMID 11228853
- [Background] Nielsen JC, Kristensen L, Pedersen AK, Mortensen PT, Pedersen OL. Changes in left atrial size and left ventricular size and functioning during follow-up of 177 patients with sick sinus syndrome randomised to atrial or dual chamber pacing. PACE 2001; 24: 697 Abstract 633
- [Background] Nielsen JC, Kristensen L, Andersen HR, Mortensen PT, Pedersen OL, Pedersen AK. A randomized comparison of atrial and dual-chamber pacing in 177 consecutive patients with sick sinus syndrome: echocardiographic and clinical outcome. J Am Coll Cardiol. 2003 Aug 20;42(4):614-23. doi: 10.1016/s0735-1097(03)00757-5. PMID 12932590
- [Background] Prech M, Grygier M, Mitkowski P, Stanek K, Skorupski W, Moszynska B, Zerbe F, Cieslinski A. Effect of restoration of AV synchrony on stroke volume, exercise capacity, and quality-of-life: can we predict the beneficial effect of a pacemaker upgrade? Pacing Clin Electrophysiol. 2001 Mar;24(3):302-7. doi: 10.1046/j.1460-9592.2001.t01-1-00302.x. PMID 11310298
- [Background] Rosenqvist M, Brandt J, Schuller H. Long-term pacing in sinus node disease: effects of stimulation mode on cardiovascular morbidity and mortality. Am Heart J. 1988 Jul;116(1 Pt 1):16-22. doi: 10.1016/0002-8703(88)90244-x. PMID 3394616
- [Background] Rosenqvist M, Bergfeldt L, Haga Y, Ryden J, Ryden L, Owall A. The effect of ventricular activation sequence on cardiac performance during pacing. Pacing Clin Electrophysiol. 1996 Sep;19(9):1279-86. doi: 10.1111/j.1540-8159.1996.tb04205.x. PMID 8880791
- [Background] Santini M, Alexidou G, Ansalone G, Cacciatore G, Cini R, Turitto G. Relation of prognosis in sick sinus syndrome to age, conduction defects and modes of permanent cardiac pacing. Am J Cardiol. 1990 Mar 15;65(11):729-35. doi: 10.1016/0002-9149(90)91379-k. PMID 2316455
- [Background] Stangl K, Seitz K, Wirtzfeld A, Alt E, Blomer H. Differences between atrial single chamber pacing (AAI) and ventricular single chamber pacing (VVI) with respect to prognosis and antiarrhythmic effect in patients with sick sinus syndrome. Pacing Clin Electrophysiol. 1990 Dec;13(12 Pt 2):2080-5. doi: 10.1111/j.1540-8159.1990.tb06946.x. PMID 1704597
- [Background] Stierle U, Kruger D, Vincent AM, Mitusch R, Giannitsis E, Wiegand U, Potratz J. An optimized AV delay algorithm for patients with intermittent atrioventricular conduction. Pacing Clin Electrophysiol. 1998 May;21(5):1035-43. doi: 10.1111/j.1540-8159.1998.tb00149.x. PMID 9604235
- [Background] Sulke N, Chambers J, Dritsas A, Sowton E. A randomized double-blind crossover comparison of four rate-responsive pacing modes. J Am Coll Cardiol. 1991 Mar 1;17(3):696-706. doi: 10.1016/s0735-1097(10)80186-x. PMID 1993790
- [Background] Sutton R, Kenny RA. The natural history of sick sinus syndrome. Pacing Clin Electrophysiol. 1986 Nov;9(6):1110-4. doi: 10.1111/j.1540-8159.1986.tb06678.x. PMID 2432517
- [Background] Toff WD, Skehan JD, De Bono DP, Camm AJ. The United Kingdom pacing and cardiovascular events (UKPACE) trial. United Kingdom Pacing and Cardiovascular Events. Heart. 1997 Sep;78(3):221-3. doi: 10.1136/hrt.78.3.221. No abstract available. PMID 9391280
- [Background] Vardas PE, Simantirakis EN, Parthenakis FI, Chrysostomakis SI, Skalidis EI, Zuridakis EG. AAIR versus DDDR pacing in patients with impaired sinus node chronotropy: an echocardiographic and cardiopulmonary study. Pacing Clin Electrophysiol. 1997 Jul;20(7):1762-8. doi: 10.1111/j.1540-8159.1997.tb03564.x. PMID 9249829
- [Background] Woodend K, Tang SI, Irvine J, Connolly S, Lav C, Paquette M, Newman D. Pacemaker dependency conditions the QOL benefits of physiologic over VVI pacing: Canadian Trial of Physiologic Pacing (CTOPP). Circulation 1999; 100(suppl I): I-20